CLINICAL TRIAL: NCT05132556
Title: The Influence of Beetroot Juice on Racial Disparities in Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Southern University (Other)
Responsible Party: Principal Investigator, Gregory Grosicki, Assistant Professor, Georgia Southern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H22040
Record Dates: First submitted 2021-11-05; First posted 2021-11-24 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Blood Pressure; Racial Disparities; Cardiovascular Risk Factor
Keywords: blood pressure; arterial stiffness; cardiovascular health; nitric oxide

STUDY DESIGN:
Intervention Model Description: The intervention is to provide participants with either nitrate-rich (~12.8 mmol nitrate; 140 mL) beetroot juice or an indistinguishable equal volume placebo with nitrate removed, the order of which will be randomized.
Who Masked: Investigator
Masking Description: The experimenter will be blinded to what condition the participant is in, and all data analysis will be conducted blinded to the condition as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (~12.8 mmol) (Experimental): Participants will have blood pressure, arterial stiffness, and blood samples (from venipuncture) assessed before and after the nitrate-rich beetroot juice (~12.8 mmol).
  Interventions: Other: Acute Beetroot Juice
- Beetroot juice with nitrate removed (Placebo Comparator): Participants will have blood pressure, arterial stiffness, and blood samples (from venipuncture) assessed before and after the beetroot juice with nitrate removed.
  Interventions: Other: Acute Beetroot Juice

INTERVENTIONS:
Other: Acute Beetroot Juice — Participants will ingest a beetroot juice supplement with and without inorganic nitrate to determine the effects of acute dietary nitrate ingestion on blood pressure and arterial stiffness

SUMMARY:
Black adults are 30% more likely to die from cardiovascular disease (CVD) compared to White adults, and more than half of this racial disparity in cardiovascular mortality may be attributed to the substantially greater prevalence of high blood pressure and vascular dysfunction in Black adults. Nitric oxide (NO) is a potent signaling molecule and key regular of vascular function that is suspected to be reduced in black individuals, but can be enriched by dietary nitrate (e.g., arugula, spinach, beets). The purpose of this study is to test the hypothesis that increasing NO bioavailability via nitrate-rich beetroot juice (BRJ) will lower blood pressure and improve vascular health in Black adults.

DETAILED DESCRIPTION:
The investigators long-term research goal is to investigate mechanisms accounting for the higher prevalence of CVD and high blood pressure in Black individuals, and identify effective preventive strategies. Nitric oxide (NO) is a gaseous molecule that plays an essential role in the regulation of vascular tone and blood pressure regulation. Some, but not all, studies have observed reduced NO bioavailability in Black individuals, which may contribute to racial disparities in vascular health. Dietary nitrate supplementation using beetroot juice (BRJ) is demonstrated to increase circulating NO, lower blood pressure and arterial stiffness, and improve blood pressure regulation in clinical populations and health individuals. The central hypothesis is that increasing NO bioavailability by nitrate-rich BRJ supplementation will lower blood pressure and improve vascular health in Black adults. The investigators acknowledge that racial differences are not entirely driven by ancestry, and thus will assess and account for sociocultural factors and health behaviors (i.e., sleep, physical activity, and nutrition) that may contribute to racial health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-39 years of age
* Body mass index (BMI) below 30 kg/m^2
* Free from signs or symptoms of neurologic, cardiovascular (e.g., heart attack, stroke, heart failure, arrhythmia), metabolic, and/or renal disease
* Have a blood pressure no lower than 90/50 mmHg
* Are not currently smoking, using smokeless tobacco, nor smoked within the past 12 months

Exclusion Criteria:

* Low blood pressure - less than 90/50 mmHg
* History of cardiovascular disease
* History of cancer
* History of diabetes
* History of kidney disease
* Obesity (BMI > 30 kg/m^2)
* Smoking or tobacco use
* Current pregnancy
* Nursing mothers
* Communication barriers

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Changes in nitric oxide (NO) metabolites | Baseline and two hours after beetroot juice ingestion, both conditions (experimental and control)
  The investigators will use chemiluminescence detection to measure salivary and circulating NO metabolites (nitrate and nitrate).
Changes in blood pressure | Baseline and two hours after beetroot juice ingestion, both conditions (experimental and control)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA), which will provide brachial and aortic blood pressures (mmHg).
Changes in arterial stiffness | Baseline and two hours after beetroot juice ingestion, both conditions (experimental and control)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV). A high-fidelity strain-gauge transducer is used to obtain the pressure waveform at the carotid pulse. Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded. PWV will be expressed as m/s.
Changes in blood pressure responses to stress | Baseline and two hours after beetroot juice ingestion, both conditions (experimental and control)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) at rest and during handgrip exercise and after exercise during cuff occlusion.
Changes in arterial stiffness responses to stress | Baseline and two hours after beetroot juice ingestion, both conditions (experimental and control)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV) at rest and during handgrip exercise and after exercise during cuff occlusion.

SECONDARY OUTCOMES:
Objective sleep duration | Baseline (pre-intervention)
  ActiGraph GT9X accelerometers will be used to quantify sleep duration. Participants will wear the watch unit for 7 days. The investigators will assess qualitative sleep scores and cross-check actigraphy wear times with a sleep diary.
Subjective sleep quality | Baseline (pre-intervention)
  The investigators will use the Pittsburgh Sleep Quality Index (0-21, higher value indicating worse sleep) to assess subjective indices of sleep health.
Physical activity | Baseline (pre-intervention)
  Participants will wear an ActiGraph GT9X accelerometer for seven days to objectively quantify time spent in moderate-vigorous physical activity.
Habitual dietary intake | Baseline (pre-intervention)
  The investigators will instruct participants to complete a diet log for three days which will be characterized with Nutrition Data System for Research (NSDR).
Social determinants of health | Baseline (pre-intervention)
  The investigators will use the Perceived Ethic Discrimination Questionnaire (22-154, higher value indicating more experiences of ethnic discrimination/racism) to quantify social determinants of health.
Economic determinants of health | Baseline (pre-intervention)
  The investigators will use the Socioeconomic Status (0-32, lower score indicating lower socioeconomic status) questionnaire to quantify economic determinants of health.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Grosicki, PhD, Principal Investigator — Georgia Southern University
Locations (1):
- Biodynamics and Human Performance Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate DMDA approvals
Supporting Information: SAP
Time Frame: One year after completion of trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of a DMDA and MTA (if needed) with Georgia Southern University and the study PI.